CLINICAL TRIAL: NCT04465500
Title: Prospective Trial of Combination External Beam Radiation Therapy and MRI-guided, Dose-differentiated High Dose-rate Prostate Brachytherapy Boost for Unfavorable-intermediate, High, and Very High-risk Prostate Cancer
Brief Title: EBRT and HDR Brachytherapy for Unfavorable-intermediate, High, and Very High-risk Prostate Cancer
Acronym: Prostate005
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Christopher Luminais, MD, Assistant Professor of Radiation Oncology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR200113
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma
Keywords: Radiation; Brachytherapy; External beam radiation therapy; Androgen Deprivation Therapy; ADT; EBRT; HDR brachytherapy; prostate cancer; MRI guided brachytherapy; brachytherapy boost
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Androgen Deprivation Therapy (ADT) High-dose-rate (HDR) Brachytherapy External Beam Radiation Therapy (EBRT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Other)
  Interventions: Radiation: External Beam Radiation; Radiation: HDR Brachytherapy; Drug: Androgen Deprivation Therapy

INTERVENTIONS:
Radiation: External Beam Radiation — EBRT will be administered every 5 consecutive days for 5 consecutive weeks. This is standard of care practice for this therapy. This may be revised as applicable per treating physician discretion. The dose of radiation will be in accordance with standard clinical practice guidelines for the treatment of prostate cancer.
  Other Names: EBRT
Radiation: HDR Brachytherapy — HDR brachytherapy will be administered per standard clinical practice (per NCCN guidelines version 1.2020 for prostate cancer), however standard clinical practice may vary between clinicians. Therefore, the dose of 15Gy in 1 fraction and a set of dosimetry guidelines are to be followed for the purposes of this study. A diagnostic MRI will be co-registered with Transrectal Ultrasound (TRUS) to perform the HDR brachytherapy.
Drug: Androgen Deprivation Therapy — The dosing and administration of ADT will be in accordance with the drug label for the drug(s) used for this purpose. Participants may receive ADT before and/or during the course of this study.
  Other Names: ADT

SUMMARY:
This study is trying to find out if the combination of Androgen deprivation therapy (ADT), MRI guided high dose radiation (HDR) brachytherapy treatment (internal radiation implant procedure) and external beam radiation therapy (EBRT) treatments lead to less side effects. This study is also looking at patient outcomes, quality of life, and overall survival for patients receiving this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male, aged 18 or above.
4. Histologic proven diagnosis of cancer of the prostate up to one year before registration.
5. Unfavorable-intermediate risk, high risk, or very high-risk prostate cancer as determined by the NCCN Guidelines Version 4.2019 (Section 12.4).
6. History and physical exam completed up to 6 months before registration.
7. PSA value < 50 ng/mL prior to androgen deprivation therapy and up to 12 months before registration. Subjects who do not meet this criteria's timeframe due to extenuating circumstances (i.e. COVID-19 quarantine, changes to their treatment plan, etc) but meet all other eligibility criteria may still be eligible. The PI will review each case and decide
8. ECOG performance status 0 or 1.
9. Pelvic MRI obtained up to 12 months before registration.
10. Candidate for receiving the combination of HDR brachytherapy and EBRT, with or without ADT. The ADT may have begun prior to study enrollment.

Exclusion Criteria:

1. Evidence of bone metastases.
2. Diagnosis of a prior invasive malignancy (except for non-melanoma skin cancer), unless the participant has been disease-free for at least 3 years.
3. Patient has had previous radical surgery (prostatectomy) or cryosurgery for prostate cancer.
4. Patient has had previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy.
5. Patient has had prior radiotherapy, including brachytherapy, to the region of this study cancer that would result in overlap of radiation therapy fields.
6. Patient has had previous or concurrent cytotoxic chemotherapy for prostate cancer (prior chemotherapy for different cancer is allowed).
7. Patient has MRI incompatible metallic implant(s) that cannot be removed.
8. The patient has severe or active co-morbidities as defined by the following:

   * Unstable angina and/or congestive heart failure requiring hospitalization up to 6 months (180 days) before registration
   * Transmural myocardial infarction up to 6 months (180 days) before registration
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * Hepatic insufficiency resulting in clinical jaundice and/or coagulation effects or severe liver dysfunction.
   * Acquired immune deficiency syndrome (AIDS) based upon current CDC definition. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be slightly immunosuppressive. Protocol- specific requirements may also exclude immuno-compromised patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Compare GU toxicity rate to the rate published in the ASCENDE-RT trial | 2 years
  Grade 3 GU toxicity rate as measured by CTCAE v5.0

SECONDARY OUTCOMES:
Estimate the prevalence of grade 3 or greater GU toxicity | 2 years
  Greater than or equal to grade 3 GU toxicity rate as measured by CTCAE v5.0
Estimate GI and sexual toxicity | 2 years
  GI and sexual toxicity as measured by CTCAE v5.0 and EPIC-26 survey results
Estimate freedom from biochemical failure (RFS) | 5 years
  Prostate-specific antigen (PSA) failure (nadir greater than 2ng/mL)
Estimate rate of undetectable PSA levels | 5 years
  PSA less than or equal to 0.2ng/mL
Describe impact of treatment on quality of life | 2 years
  EPIC-26 survey results

CONTACTS AND LOCATIONS:
Overall Officials: Chris Luminais, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States